CLINICAL TRIAL: NCT00120068
Title: Improving Care for Nursing Home Pneumonia in NHCUs and Veterans' Homes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Masking: None | Purpose: Prevention
Other Study IDs: IIR 03-123
Record Dates: First submitted 2005-07-01; First posted 2005-07-14 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Concurrent Review

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Nursing inservices; Procedure: Academic detailing to MDs; concurrent review and feedback

INTERVENTIONS:
Behavioral: Nursing inservices
Procedure: Academic detailing to MDs; concurrent review and feedback

SUMMARY:
Nursing Home Acquired Pneumonia (NHAP) causes excessive morbidity, mortality, hospitalization, and loss of function. At any given time, 1.1-2.5% of veterans who reside at nursing home care units (NHCUs) and State Veterans Homes (SVHs) are ill with pneumonia. Multi-faceted implementation of evidence-based guidelines has been shown to be feasible in the private sector. Retrospective studies demonstrate an association between guideline adherence and improved survival.

DETAILED DESCRIPTION:
Background:

Nursing Home Acquired Pneumonia (NHAP) causes excessive morbidity, mortality, hospitalization, and loss of function. At any given time, 1.1-2.5% of veterans who reside at nursing home care units (NHCUs) and State Veterans Homes (SVHs) are ill with pneumonia. Multi-faceted implementation of evidence-based guidelines has been shown to be feasible in the private sector. Retrospective studies demonstrate an association between guideline adherence and improved survival.

Objectives:

Assess the feasibility of a QUERI-like strategy to translate the guidelines into practice at VA-affiliated nursing homes through focus groups, interviews, and a small intervention trial.

Methods:

Nursing staff focus groups, key informant interviews, and tests of academic detailing (educational outreach) scripts were conducted at five facilities. Based on the information gathered, the QUERI-like intervention was modified and tested at the Florence, Colorado SVH during one influenza season compared to no intervention at a nearby SVH. Forty random SVH nursing staff took an anonymous telephone survey of knowledge and attitudes about NHAP twice prior to the intervention. A second randomly selected group of CNAs and nurses took the survey after the intervention. Research assistants enrolled residents with NHAP, interviewed them and their nurses about their quality of life, assessed their function and reviewed their medical records. The intervention was multifaceted, including (1) a formative phase to tailor implementation and foster staff investment in process and outcomes, (2) institutional level change to facilitate immunization and use of appropriate antibiotics and tests; (3) interactive educational sessions to improve nursing assessment; and (4) academic detailing to physicians to impact diagnostic and prescribing practices. Data were analyzed by Template Analysis Technique for qualitative data; test-retest reliability of the knowledge and attitude survey; exploratory bivariate comparison of intervention delivery and uptake, process of care and outcomes between the intervention and control facilities.

Status:

Project work is ongoing.

ELIGIBILITY:
Inclusion Criteria:

Residents of Florence and Walsenburg, Colorado State Veterans Homes

Exclusion Criteria:

Residents within 48 hours of death or if in facility < 5 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-11; Primary Completion 2005-03 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn A. Hutt, MD, Principal Investigator — VA Eastern Colorado Health Care System, Denver, CO
Locations (1):
- VA Eastern Colorado Health Care System, Denver, CO, Denver, District of Columbia, United States

REFERENCES:
- [Result] Levy C, Hutt E, Pointer L. Site of death among veterans living in Veterans Affairs nursing homes. J Am Med Dir Assoc. 2012 Mar;13(3):199-201. doi: 10.1016/j.jamda.2011.08.004. Epub 2011 Sep 25. PMID 21945536
- [Result] Hutt E, Ruscin JM, Corbett K, Radcliff TA, Kramer AM, Williams EM, Liebrecht D, Klenke W, Hartmann S. A multifaceted intervention to implement guidelines improved treatment of nursing home-acquired pneumonia in a state veterans home. J Am Geriatr Soc. 2006 Nov;54(11):1694-700. doi: 10.1111/j.1532-5415.2006.00937.x. PMID 17087696